CLINICAL TRIAL: NCT06376981
Title: Benefit of a Subacromial Injection Combining Corticosteroid and Hyaluronic Acid Versus Corticosteroid Alone in Supraspinatus Tendinopathy
Brief Title: Hyaluronic Acid in Shoulder Tendinopathy
Acronym: ACCTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHD23_0025
Record Dates: First submitted 2024-04-11; First posted 2024-04-22 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Shoulder Tendinitis
Keywords: Shoulder tendinitis; Hyaluronic acid; Corticosteroid injection
MeSH Terms: interventions — Hyaluronic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination of corticosteroid and hyaluronic acid injection (Experimental): An injection of 1 ml if corticosteroids and an injection of 2 ml of hyaluronic acid
  Interventions: Drug: Hyaluronic acid injection; Drug: Corticosteroid injection
- Corticosteroid injection alone (Placebo Comparator): An injection of 1 ml of corticosteroids and an injection of 2 ml of placebo (physiological serum).
  Interventions: Drug: Corticosteroid injection; Drug: Placebo injection

INTERVENTIONS:
Drug: Hyaluronic acid injection — An injection of 2 ml of Acid hyaluronic
  Arms: Combination of corticosteroid and hyaluronic acid injection
Drug: Corticosteroid injection — An injection of 1 ml of corticosteroids
Drug: Placebo injection — An injection of 2 ml of placebo (physiological serum)
  Arms: Corticosteroid injection alone

SUMMARY:
Multicentric, randomised study to compare the effectiveness on activity pain at 3 months of corticosteroid injection associated with hyaluronic acid with corticosteroids injection alone in patients with tendinopathy of the supraspinatus with clinical reevaluation at one, three and six months.

ELIGIBILITY:
Inclusion Criteria:

* Active patient aged between 18 and 65;
* Patient suffering from pain compatible with supraspinatus tendinopathy for at least 2 months;
* Patient with simple tendinopathy or partial tendon rupture;
* Patient with tendinopathy confirmed by ultrasound or MRI;
* Patient with an active pain visual analog scale ≥ 4 for more than 6 weeks;
* Patient with an active pain visual analog scale ≥ 4 on the day of inclusion;
* Patient failing medical treatment (rest, analgesics, NSAIDs, physiotherapy);
* Patient able to follow the protocol and having given oral informed consent to take part in the research;
* Patient affiliated to the social security system or entitled person;

Exclusion Criteria:

* Patient suffering from a transfixing tendon rupture;
* Patients suffering from post-traumatic tendon rupture;
* Patients suffering from calcific tendinopathy (calcification > 5 mm);
* Patients with associated glenohumeral osteoarthritis;
* Patients with associated symptomatic acromioclavicular osteoarthritis;
* Patients with shoulder pain for reasons other than tendinopathy (capsulitis, chronic inflammatory rheumatism, fibromyalgia, amyloidosis);
* Patients who have had a subacromial infiltration in the previous 6 months;
* Patients with a known allergy to one of the products including their excipients (methyl parahydroxybenzoate, propyl parahydroxybenzoate, benzyl alcohol);
* Patients with a known allergy to lidocaine;
* Patients with a local or generalised infection, or suspected infection;
* Patients with severe coagulation disorders or taking anticoagulants;
* Patients with severe and/or uncontrolled hypertension > 160/100 mmHg;
* Patients with unbalanced diabetes (last HbA1c > 8.5%);
* Patients with a history of addiction to psychoactive substances;
* Patient participating in another clinical research protocol with an impact on the research objectives;
* Patient already randomised in the study;
* Patient who is pregnant, parturient, breastfeeding or able to procreate without effective contraception* in the month prior to inclusion and up to 15 days after infiltration;
* Patients under guardianship, curators or deprived of liberty;
* Patient under a mandate for future protection activated ;
* Patient under family guardianship ;
* Patient under court protection ;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale pain on activity ranging from 0 to 100 mm at month 3. | Month 3
  Visual analog scale pain on activity ranging from 0 to 100 mm at month 3. Pain is defined by the worst pain felt during active examination: anterior elevation, abduction, internal and external rotation, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Céline COZIC, Dr, Principal Investigator — Centre Hospitalier Départemental Vendée
Locations (2):
- France (2):
  - CHD Vendée, La Roche-sur-Yon
  - CHU Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No